CLINICAL TRIAL: NCT05975190
Title: Respiratory Training and Relaxation Techniques to Improve Adjuvant Radiation Therapy in DIBH in Breast Cancer Patients - B-REST-Study
Brief Title: Respiratory Training and Relaxation Techniques to Improve Adjuvant Radiation Therapy in DIBH in Breast Cancer
Acronym: B-REST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: German Cancer Aid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-277_1-S-NP
Record Dates: First submitted 2023-07-12; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-01

CONDITIONS: Radiotherapy; Breast Cancer; Relaxation; Breathholding
Keywords: Adjuvant radiotherapy for Breast Cancer; DIBH in left sided Breast Cancer; Respiratory and Relaxation Techniques; patients compliance; active participation under radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The randomized design of the study will test R&R interventions compared to current conventional DIBH instruction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R&R arm (interventional arm) (Experimental): The training program in the experimental arm includes relaxation techniques, breath hold training, music, and nature sounds that patients can listen to on an MP3 player. The training is offered one week before the planning CT scan and patients are encouraged to practice independently. Patients complete standardized questionnaires about their well-being and satisfaction at prospective time points before, during the radiation treatment course, as well as at 6 weeks follow-up.
  Interventions: Other: Respiratory training and relaxation techniques under adjuvant radiation therapy in DIBH in breast cancer
- Standard arm (No Intervention): Patients in the standard arm receive current conventional DIBH instruction without an extended R&R training. Patients complete standardized questionnaires about their well-being and satisfaction at prospective time points before, during the radiation treatment course, as well as at 6 weeks follow-up.

INTERVENTIONS:
Other: Respiratory training and relaxation techniques under adjuvant radiation therapy in DIBH in breast cancer — R&R training provided on an MP3-player for daily practice
  Arms: R&R arm (interventional arm)

SUMMARY:
The goal of this prospective clinical trial is to improve patient compliance and performance of deep inspiration breath hold (DIBH) to further reduce the cardiac dose from left breast radiation, and to improve cooperation and patient satisfaction through an active and formal pre-treatment respiratory training program combined with relaxation training (R&R) in breast cancer patients undergoing adjuvant radiotherapy for left sided breast cancer.

The main questions the study aims to answer are:

* Does the use of communication training and the use of relaxation techniques (R&R) reduce the Maximum dose to the heart (Dmax) and improve further heart dose parameters in deep inspiration during adjuvant radiotherapy for breast cancer?
* Does R&R improve longitudinal anxiety and quality of life under patients undergoing DIBH adjuvant radiotherapy for left sided breast cancer?

Participants will be randomly assigned to either an experimental arm, which will receive the R&R, versus a standard arm that will not receive the R&R.

* training program in the experimental arm includes breath hold training, music, and nature sounds that patients can listen to on an MP3 player
* both groups complete standardized questionnaires about their well-being and satisfaction at prospective time points before, during the radiation treatment course, as well as at 6 weeks follow-up

Researchers will compare the R&R group (interventional arm) to current conventional DIBH instruction (standard group) to see if Dmax to the heart decreases and compliance and satisfaction under patients rises.

DETAILED DESCRIPTION:
Postoperative radiotherapy is widely practiced and highly effective in enabling breast conserving therapy in early stage tumors, and decreasing recurrence while improving survival in patients with advanced-stage breast cancer, the most common cancer in women. However, these benefits of radiotherapy are associated with a long-term risk of cardiac morbidity and mortality in breast cancer survivors. The unintended cardiac radiation exposure due to the heart's proximity to the treatment target has been well recognized, particularly in left-sided breast cancer. Because there is no lowest "safe" threshold radiation dose level for radiation-induced cardiac complications, the dose to the heart must be kept as low as possible to reduce the complications risk.

Recent advances in high-precision 3D conformal and intensity-modulated radiotherapy techniques have enabled better protection of the heart. Treatment in deep inspiration breath hold (DIBH) is indispensable to realize these technological capabilities by taking advantage of the greater distance created between the radiotherapy target and the contralaterally and inferiorly displaced heart during deep inspiration. While many studies have demonstrated reduction of the heart dose with DIBH, challenges in decreasing heart dose to a minimum remain.

Radiotherapy in DIBH requires active and complex cooperation from the patient, and its success critically depends on how well patients are capable to perform the prolonged extended deep breathing maneuver on a repetitive basis every day during their weeks-long treatment course. Both the physical demands and profound anxiety and stress, which are highly prevalent in breast cancer patients, additionally interfere with patients' DIBH performance. Anxiety is well known to directly adversely affect breathing patterns, thereby challenging patients' ability to perform DIBH optimally.

Preliminary research explored the role of physical training and showed that targeted DIBH training improves patients' cooperation and the ease of the DIBH procedure, and reduces the radiation dose to the heart. However, while DIBH training regimens may improve patients' physical respiratory skill levels, they do not address their mental stress and anxiety. Relaxation techniques to alleviate anxiety and stress have been rarely used in complex radiotherapy procedures, particularly not in DIBH. Preliminary studies in diagnostic radiology procedures suggest that advanced communication and relaxation techniques, targeted to relieve anxiety and stress, improve patients' procedural performance, anxiety and comfort. The investigators hypothesize that implementing both, DIBH Respiratory Training and advanced communication and Relaxation Training (R&R), improve patients' DIBH performance skills and further reduce heart dose, while alleviating anxiety and stress and improving quality of life during and after radiation therapy.

The investigators propose to test this hypothesis in a clinical trial randomizing R&R vs. standard-of-care management in patients with radiotherapy in DIBH for left breast cancer. The investigators primary endpoint will assess heart dose (Dmax), and secondary endpoints include longitudinal anxiety and quality of life assessment and clinic workflow efficiency. The ultimate goal of this proposal is to develop a validated patient-centered training and integrative health regimen to further improve the success of advanced-technology-based cardiac dose reduction, and improve cardiac health in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients
* Left sided breast cancer
* Treated with surgery prior to radiotherapy
* Age >18 years at time of inclusion
* WHO performance status 0-1
* Planned for radiotherapy alone to the breast, the chest wall and/or the lymph node areas
* Radiotherapy based on planning-CT scan using either 3D-CRT, IMRT, or VMAT/RapidArc
* Written Informed consent

Exclusion Criteria:

* Age <18 years
* Pregnancy, Breastfeeding
* Previous thoracic or mediastinal radiation
* Bilateral breast cancer
* Partial breast irradiation
* M1 disease (metastatic breast cancer)
* Severe lung disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 108 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Dmax to the heart in DIBH under adjuvant radiotherapy of left sided breast cancer | during treatment (4 weeks)
  Maximum Dose to the heart (Dmax) in deep inspiration during adjuvant radiotherapy for breast cancer in dependence of the use of communication training and the use of relaxation techniques

SECONDARY OUTCOMES:
Improving quality of life under radiotherapy of left sided breast cancer | - at baseline - during treatment (4 weeks) - at 6 week Follow-Up
  Quality of life outcome measures using a standardized questionnaire including parts of EORTC- Quality of Life-C30 (high score for a functional scale or global health status represent a high level of functioning or a high QoL, a high score for a symptom scale represents a high level of problems; scale: 0 - 100)
Improving heart Dmean under radiotherapy of left sided breast cancer | during treatment (4 weeks)
  Change in heart Dmean as a measure of cardiac toxicity
Improving Left anterior descending (LAD) Dmean under radiotherapy of left sided breast cancer | during treatment (4 weeks)
  Change in LAD Dmean as a measure of cardiac toxicity
Improving LAD Dmax under radiotherapy of left sided breast cancer | during treatment (4 weeks)
  Change in LAD Dmax as a measure of cardiac toxicity
Improving left ventricle (LV) Dmean under radiotherapy of left sided breast cancer | during treatment (4 weeks)
  Change in LV Dmean as a measure of cardiac toxicity
Evaluation of clinic workflow metrics under radiotherapy of left sided breast cancer | - before start of treatment (one week before planning CT) - during treatment (4 weeks) - at 6 week Follow-Up
  Evaluation of clinic workflow metrics in the radiation oncology unit related to the implementation of DIBH by measuring specific data, such as total treatment time, in comparison with metrics of patients in the control group.
Improving patients satisfaction with R&R under radiotherapy of left sided breast cancer | - during treatment (4 weeks) - at 6 week Follow-Up
  Patient-reported outcome measures using a standardized questionnaire including parts of EORTC-Qualitiy of Life-BR-23 (Breast Cancer score, higher scores mean a worse outcome; scale: 0-100)
Improving radiation dose in organs at risk under radiotherapy of left sided breast cancer | during treatment (4 weeks)
  Comparison of radiation doses in organs at risk of structures other than the heart as a criterion for sparing adjacent organs and structures

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Combs, MD, Principal Investigator — Department of Radiation Oncology, Technical University of Munich
Locations (1):
- Department of Radiation Oncology, Technical University of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: No